CLINICAL TRIAL: NCT03349203
Title: Icotinib as Neoadjuvant and Adjuvant Therapy in EGFR-mutant Stage IIIB or Oligometastasis Non-small Cell Lung Cancer: a Single Arm, Phase II Clinical Study
Brief Title: Icotinib as Neoadjuvant and Adjuvant Therapy in EGFR-mutant Stage IIIB or Oligometastasis Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV81
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-01

CONDITIONS: EGF-R Positive Non-Small Cell Lung Cancer
MeSH Terms: interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icotinib (Experimental): Patients with EGFR-mutant stage IIIB or oligometastasis Non-small Cell Lung Cancer which can be potentially radical treated by surgery are arranged to receive Icotinib with a dose of 125 mg three times per day orally for 8 weeks before surgery and 2 years as adjuvant therapy after surgery or till progressive disease or unaccepted toxicity.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Patients with EGFR-mutant stage IIIB or oligometastasis Non-small Cell Lung Cancer which can be potentially radical treated by surgery are arranged to receive Icotinib with a dose of 125 mg three times per day by mouth for 8 weeks as neoadjuvant therapy before surgery and 2 years as adjuvant therapy or till progressive disease or unaccepted toxicity.
  Other Names: Conmana

SUMMARY:
The main purpose of this study is to evaluate the pulmonary and metastases lesions objective response rate after Icotinib preoperative therapy in EGFR-mutant stage IIIB or oligometastasis Non-small Cell Lung Cancer which can be potentially radical treated by surgery.

DETAILED DESCRIPTION:
Patients with EGFR-mutant stage IIIB or oligometastasis Non-small Cell Lung Cancer which can be potentially radical treated by surgery are arranged to receive Icotinib with a dose of 125 mg three times per day orally for 8 weeks as neoadjuvant therapy; then they receive surgical resection of the tumor. If there is curative effect of Icotinib according to the RECIST or pathological report, the patients will continue receive Icotinib for two years as adjuvant therapy after surgery or till progressive disease or unaccepted toxicity. The primary objective of this study is evaluate the pulmonary and metastases lesions objective response rate after Icotinib preoperative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histology or cytology confirmed Non-small Cell Lung Cancer; EGFR mutation (EGFR 19del and/or 21L858R) detected by tumor tissue biopsy of primary lesion or metastatic lesion or plasma ctDNA
* No previous anti-tumor treatment such as surgery, chemotherapy, radiotherapy or biological therapy
* Stage IIIB or IV Oligometastasis Non-small Cell Lung Cancer. (a) stage IV Oligometastasis: the metastasis organ mainly include: 1. adrenal metastasis which can be potentially resected by surgery or radically treated by SRS radiotherapy; 2. brain metastasis which can be potentially resected by surgery or radically treated by SRS radiotherapy. At the same time, the primary lesion of the lung can be completely removed, which should be T1-2, N0-1 or T3, N0. (b) stage IIIB (T1-3, N3): it is limited to patients who are unsuitable or refuse to accept pulmonary primary lesion radiotherapy. It only include subclavian lymph node or anterior scalenus lymph node metastasis (mediastinal lymph node metastasis is excluded by PET-CT). The metastasis lesion should be single or less than 3, its diameter is no more than 3 cm and can be potentially resected.
* Sufficient tumor histological specimens (non-cytology) for molecular marker analysis
* At least one lesion with measurable diameter and its longest diameter is large than 10 mm by CT measurement

Exclusion Criteria:

* Previous systemic anti-tumor treatment of Non-small Cell Lung Cancer, including cytotoxic drug therapy, targeted drug therapy (tyrosine kinase inhibitors or monoclonal antibodies) and experimental treatment, etc
* Previous local radiotherapy of Non-small Cell Lung Cancer
* Be allergic to any component of Icotinib tablet (Conmana)
* Other cancers within five years prior to the treatment of this study. Except for cervical carcinoma, basal cell carcinoma and bladder epithelial neoplasm (including Ta and Tis)
* Any instable systemic disease, including: active infection, high blood pressure out of control, unstable angina, onset of angina pectoris within the past 3 months, congestive heart failure, myocardial infarction, severe arrhythmia, liver, kidney or metabolic disease
* Previous interstitial lung disease, drug-induced interstitial disease, radiation pneumonia requiring hormone therapy or any active intersexual lung disease with clinical evidence
* Idiopathic pulmonary fibrosis detected by CT scan at baseline;
* Not fully controlled eye inflammation or infections, or any condition that may lead to the above eye diseases
* Human immunodeficiency virus infection
* Patients undergoing major surgery or severe trauma within 2 months prior to the first use of the experimental drug
* Patients with Small Cell Lung Cancer
* Pregnant or lactating women
* Neurological or psychiatric disorders history, including epilepsy or dementia
* Other situations not appropriate to enter the group considering by the investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate as assessed by RECIST1.1 | eight weeks
  Objective Response Rate was defined as the percentage of participants whose tumor lesions disappear completely or diameters reduced by at least 30% as assessed by RECIST1.1.

SECONDARY OUTCOMES:
Disease Control Rate as assessed by RECIST1.1 | five years after surgery
  Disease Control Rate was defined as the total percentage of participants except for those with tumor lesions diameters increased by at least 20% as assessed by RECIST1.1.
Time to Tumor Progression as assessed by RECIST1.1 | five years after surgery
  Time to Tumor Progression was defined as the time between participants' randomization and their tumor progression as assessed by RECIST1.1.
Overall survival of participants | five years after surgery
  Overall survival was defined as the time from participants' randomization to their death due to any cause.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | five years after surgery
  The number of participants with treatment-related adverse events as assessed by CTCAE v4.0 would be recorded and calculated after them participating into the study and taking the experimental drug.

CONTACTS AND LOCATIONS:
Overall Officials: Shugeng Gao, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Science, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes